CLINICAL TRIAL: NCT01589913
Title: Remote Care for Reducing Cardiac Fear, Fear of Dying, Depression, and Increasing Quality of Life in ICD-Patients With Cardiac Insufficiency/at Risk for Fatal Cardiac Arrhythmia.
Brief Title: REmote Web Assisted Care for Heart Failure Patients With Implantable Cardioverter Defibrillators
Acronym: REACH-ICD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: University of Wuerzburg (Other); Campus Bad Neustadt (Other); Hospital Rothenburg ob der Tauber (Unknown); University Hospital Brandenburg (Unknown); Klinikum Aschaffenburg-Alzenau (Other); Klinikum Bad Woerishofen (Unknown); University of Leipzig (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UKW-CHFC-G2
Record Dates: First submitted 2011-10-05; First posted 2012-05-02 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Anxiety; Depression; Quality of Life
Keywords: Implantable Cardioverter Defibrillators; Heart Failure; Anxiety; Depression; Quality of Life; Remote Care; Prevention
MeSH Terms: conditions — Anxiety Disorders; Depression; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment as usual plus remote care (Experimental): The same treatment as described under "treatment as usual" plus participation in the intervention "ICD-Forum".
  Interventions: Behavioral: ICD-Forum
- Treatment as usual (No Intervention): Standard information provided by hospitals on ICD-technology as well as consequences of ICD-implantation plus medical aftercare including cardiology appointments at 1, 3, and 6 months, and one year after ICD-implantation.

INTERVENTIONS:
Behavioral: ICD-Forum — The CBT based internet program ICD-Forum is designed to increase QoL, and decrease anxiety and depression in ICD-patients. The program includes a therapist moderated asynchronous discussion group and content focused modules following a six weeks schedule:
  1. Introduction to participants and online system
  2. Knowledge regarding ICDs
  3. Strategies for behavior change
  4. Psychological models for anxiety and depression
  5. Strategies to cope with avoidance, anxiety and depression
  6. Resume, evaluation, resolution of open questions, goal setting, good bye
  Other Names: www.icd-forum.de; icd-forum.de; REACH-ICD
  Arms: Treatment as usual plus remote care

SUMMARY:
Aim and Background: Although implantable cardioverter defibrillators (ICD) save lives, many ICD-patients experience psychosocial complications such as anxiety disorders, depression and reduced quality of life after ICD-implantation. A recent review has indicated great potential for psychosocial interventions to reduce anxiety and to increase exercise capacity of ICD-patients. In a previous study, the investigators showed that mailed information about technical, medical and psychological effects of ICD plus phone counseling are effective interventions for reducing anxiety, psychological distress and increasing QoL in ICD-patients < 65 years. In a pilot study the investigators also documented promising effects of an internet based intervention with similar content.

Method: In a prospective, multicenter, multidisciplinary, half-open, part-randomized, controlled clinical trial N = 200 patients with an ICD will either receive medical care as usual or additionally attend a psychosocial prevention program via remote care. Psychosocial support will be provided utilizing the advantages of the internet. Thus, patient-centered support will be offered independent from time and location.

Outcome measures are psychometric data (questionnaires on cardiac fear, etc.), cardiac functioning, and clinical status which will be assessed up to 1 week before ICD-implantation (T0), in week 1 (T1) and within one week after (T2) the 6-weeks prevention program, and 12 months after T0 (T3). Furthermore, demographic data, personality characteristics, expectations, physiology, pro-inflammatory cytokines and cardiac status will be assessed as mediating or moderating variables.

Hypotheses: A web-based psychosocial intervention in addition to medical care as usual leads to increased QoL and reduced anxiety and depression. Secondary goals are the identification of psychosocial and medical predictors, mediators, and moderators of treatment efficacy. Moreover, differences between patients with ICDs implanted for primary vs. secondary prevention will be explored.

Conclusion: This project will evaluate the feasibility and efficacy of an internet based intervention for ICD-patients. Furthermore, the investigators aim at identifying predictors and mediators of treatment outcome. This will improve interdisciplinary care for ICD-patients; further applications for other cardiovascular disorders as well as preventive programs for heart failure seem possible.

DETAILED DESCRIPTION:
See Summary.

ELIGIBILITY:
Inclusion Criteria:

* Implanted ICD
* Internet access can be installed during completion of the prevention program

Exclusion Criteria:

* Medical reasons preventing participation of the prevention program (e.g. emergency hospitalization) for more than one week of the program
* Suicidality (Patients with scores > 8 on the depression subscale of the HADS will be assessed via interviews conducted by a qualified psychologist)
* Severe cognitive impairment (< 17 points in the MMST; Kessler, J., Markowitsch, H. J. & Denzler, P. (2000). Mini-Mental-Status-Test (MMST). Göttingen: Beltz Test GMBH. [Deutsche Adaption])
* Insufficient command of German to follow the intervention program
* Current ICD-10 diagnosis:
* F1x: Mental and behavioral disorders due to psychoactive substance use
* F2x: Schizophrenia, schizotypal and delusional disorders
* F30: Manic Episode
* F31: Bipolar affective disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
change of psychosocial well-being (combined score for measures of anxiety, depression, and quality of life) from week 1 (T1) to one week after (T2) the 6-weeks prevention program | up to 1 week before ICD-implantation (T0), in week 1 (T1) and within one week after (T2) the 6-weeks prevention program, and 12 months after T0 (T3)
  assessment tools for aspects of psychosocial well-being (German versions will be used): Anxiety: Cardiac Fear Questionnaire (Hoyer & Eifert, 2001); Depression: Hospital Anxiety and Depression Scale (Hinz & Brähler, 2011); QoL: MOS 36-item short-form health survey (Ware & Sherbourne, 1992)

SECONDARY OUTCOMES:
1. Health status 2. ICD-related trauma 3. Life-style factors 4. ICD-Related concerns 5. Psychological well-being 6. Type-D personality 7. Social support 8. Economic efficiency | up to 1 week before ICD-implantation (T0), in week 1 (T1) and within one week after (T2) the 6-weeks prevention program, and 12 months after T0 (T3)
  1. assessed by NYHA-class, LVEF, blood pressure
  2. measured through IES, Maercker, & Schützwohl, 1998 and PDEQ, Fuglsang, Moergeli, et al., 2002 and FSAS, Kuhl, et al., 2006
  3. measured through smoking, BMI
  4. measured through FPAS, Burns, et.al., 2005 and ICD-Safety and Concerns Scales, Crössmann, 2005
  5. measured through SCL-9-K, Klaghofer & Brähler, 2001
  6. measured through DS14, Grande, et al., 2004
  7. measured through BSSS, Schulze, & Schwarzer, 2003
  8. measured according to Schweikert, Hahmann & Leidl, 2008
psychophysiological parameters: heart rate variability | up to 1 week before ICD-implantation (T0) and 1, 3, 6, and 12 months after ICD-implantation
  time- and frequency domain parameters of HRV (Camm et al., 1996)
biometric markers: 1. proinflammatory cytokines 2. coagulation parameters | up to 1 week before ICD-implantation (T0) and 6 months after ICD-implantation
  1. ELISA analysis of IL-1β, IL-6, TNF-α
  2. Fibrinogen

CONTACTS AND LOCATIONS:
Overall Officials: Paul Pauli, Prof. Dr., Principal Investigator — University of Würzburg; Stefan M Schulz, Dr., Principal Investigator — University of Würzburg
Locations (7):
- Germany (7):
  - Department of Cardiology, Center of Cardiovascular Medicine, Bad Neustadt an der Saale, Bavaria
  - Klinik Bad Wörishofen, Bad Wörishofen, Bavaria
  - Department of Internal Medicine, Krankenhaus Rothenburg ob der Tauber, Rothenburg upon Tauber, Bavaria
  - University of Wuerzburg, Würzburg, Bavaria
  - Wuerzburg University Hospital, Department of Medicine I (Cardiology), Würzburg, Bavaria
  - Klinikum Aschaffenburg-Alzenau, Aschaffenburg, Hesse
  - Klinik für Kardiologie und Pulmologie, Medizinische Hochschule Brandenburg, Brandenburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schulz SM, Pauli P. [Internet therapy for ICD-patients]. Herzschrittmacherther Elektrophysiol. 2011 Sep;22(3):166-73. doi: 10.1007/s00399-011-0145-y. German. PMID 21826541
- [Background] Schulz SM, Massa C, Grzbiela A, Dengler W, Wiedemann G, Pauli P. Implantable cardioverter defibrillator shocks are prospective predictors of anxiety. Heart Lung. 2013 Mar-Apr;42(2):105-11. doi: 10.1016/j.hrtlng.2012.08.006. Epub 2012 Oct 27. PMID 23110854
- [Result] Schulz SM, Ritter O, Zniva R, Nordbeck P, Wacker C, Jack M, Groschup G, Deneke T, Puppe F, Ertl G, Angermann C, Stork S, Pauli P. Efficacy of a web-based intervention for improving psychosocial well-being in patients with implantable cardioverter-defibrillators: the randomized controlled ICD-FORUM trial. Eur Heart J. 2020 Mar 14;41(11):1203-1211. doi: 10.1093/eurheartj/ehz134. PMID 30957867
- See also: Homepage for ICD-Forum, the remote care program evaluated in REACH-ICD — http://www.icd-forum.de